CLINICAL TRIAL: NCT01273584
Title: Does Metformin Improve Pregnancy Outcomes (Incidence of LGA (≥90% Birth Weight Centile) Babies, Onset of Maternal GDM, Hypertension, PET, Macrosomia, Shoulder Dystocia, Admission to SCBU) in Obese Non-diabetic Women?
Brief Title: Metformin in Obese Non-diabetic Pregnant Women
Acronym: MOP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Epsom and St Helier University Hospitals NHS Trust (Other)
Collaborators: Fetal Medicine Foundation (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WCH/2008/001; 2008-005892-83 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Pregnancy Complications; Obesity
Keywords: Metformin, obese, pregnancy, gestational diabetes
MeSH Terms: conditions — Pregnancy Complications; Obesity; Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Tablet Metformin 500 mg, starting dose of 1 tablet twice a day with meals, gradually titrated upwards by 1 tablet every week to a maximum dose of 2 tablets three times a day.
  Tablets started at recruitment and continued till the delivery of the baby
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Tablet Placebo 500 mg, starting dose of 1 tablet twice a day with meals, gradually titrated upwards by 1 tablet every week to a maximum dose of 2 tablets three times a day.
  Tablets started at recruitment and continued till the delivery of the baby
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Maximum dosage 500 mg 2 tablets 3 times a day (with each meal) start with 1 tablet twice a day and gradually titrate upwards to maximum dose
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Placebo maximum dosage 2 tablets 3 times a day ( with meals) start with 1 tablet twice a day and gradually titrate upwards to maximum dose
  Other Names: Dummy tablet
  Arms: Placebo

SUMMARY:
Obesity is on the rise in all developed countries. Of particular concern is that more young people including children are being recognised as being overweight or obese. We know from a recent large national enquiry into all maternal and child deaths in the UK, known as CEMACH, that obesity is a major risk both for the mother and her child. When all deaths in women during pregnancy are analysed, obesity comes out as the most common risk factor. Babies of obese mothers are more than 3 times as likely to need admission to the Neonatal Intensive Care Unit.

Traditionally, obesity is treated by lifestyle measures encouraging healthy eating and increasing physical activity. Unfortunately these measures are often insufficient to produce significant improvements in weight. If obese women gain little or even no weight during pregnancy, the outcome of the pregnancy is known to be improved. This was shown in a very large study of more than 120, 000 obese women.

The drug metformin has been used for years in the treatment of diabetes and more recently for polycystic ovary syndrome (PCOS). Studies in pregnant PCOS women and women with diabetes in pregnancy have shown it to be safe and effective. Fortunately it is relatively cheap and taken as a tablet with meals.

Metformin has the great advantage of not causing weight gain and often leads to a small amount of weight loss. It works by improving the body's sensitivity to insulin which is important as resistance to insulin is common in obesity.

We have a lot of experience using metformin to treat women with diabetes in pregnancy where it is greatly beneficial. We now wish to examine its potential for obese women who do not have diabetes. We are hoping to show that it will benefit these women by causing less weight gain, less high blood pressure, and less diabetes. We anticipate babies will also have better birth weights, will be easier to deliver naturally, will not need to go to special care baby units and will be healthier.

DETAILED DESCRIPTION:
Obesity in Pregnancy has been identified by the Confidential Enquiry into Maternal and Child Health [CEMACH] report (2007) as a major health risk to mother and baby:

* 35% of women who died were obese
* 30% of the mothers who had a stillbirth or a neonatal death were obese

Obesity increases the risk of miscarriages, GDM, pregnancy-induced hypertension/PET, Caesarean sections, deep venous thrombosis, puerperal sepsis and LGA babies. There is a 5-fold increase in costs of antenatal care. Results from various studies have concluded that limited or no weight gain during pregnancy in obese women results in more favourable pregnancy outcomes. By improving insulin sensitivity and enhancing GLP-1 release, metformin is associated with weight reduction by approximately 5.8% with no serious adverse events.

The aim of this study is to test the hypothesis that management of obese non-diabetic pregnant women with standardised life-style intervention (diet and physical activity) plus metformin will lead to improved maternal and perinatal outcomes compared with life-style intervention alone.

The study will also seek to determine whether metformin will improve body fat distribution as measured by bioimpedance during pregnancy with particular emphasis on metabolic active visceral fat.

Genetic studies will investigate whether patients with polymorphisms of the candidate fat gene, FTO gene, differ in their response to metformin and whether this is associated with favourable pregnancy outcomes.

This is a randomised, multicentre, double blind, placebo-controlled trial.Assuming power 90%, significance level 5% and 2-sided testing, we will recruit 425 subjects per arm of the trial.This will allow the detection of a difference in mean centile (z-score) of 0.21 standard deviations.

All women will undergo oral glucose tolerance testing at booking and at 28 wks; those found to have GDM at 28 weeks will commence home glucose monitoring and will receive metformin if glucose values are outside target range.

The primary outcome will be the birth weight centile (z score). Secondary outcomes include maternal and neonatal outcomes, body composition scores, patient satisfaction and infant development at 2 years. The relation between FTO gene variants and pregnancy outcomes will be examined. Parametric and non-parametric tests will be used as appropriate.

This is a multicentre trial to be undertaken in 7 centres in the UK over a period of 3 years in order to reach the required sample size. Mr Hassan Shehata, Clinical lead and Consultant Obstetrician and Gynecologist is the Chief Investigator of the trial and the trial will be centrally coordinated by Dr Jyoti Balani at Epsom and St Helier University Hospital. In the first phase of the research, we would be recruiting a total of 546 pregnant women into the trial. 200 women would be recruited at Epsom and St Helier Hospital, 200 women at kings college Hospital under the supervision of Professor Kypros Nicolaides and 146 at Royal Surrey County Hospital under the supervision of Dr Lesley Roberts.

Given the low cost of metformin and the potentially high impact on health for both mother and baby, we anticipate the study will show metformin to be highly cost-effective. We anticipate improved patient satisfaction scores in those taking metformin as they gain less weight and develop fewer complications. Improvements in the metabolic milieu during interuterine growth is expected to improve long term outcome for the infants of mothers treated with metformin.

Benefits to patients will be immediate from the time the project's findings are presented. Implementation into clinical practice is expected to greatly benefit the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women with BMI>35
* Informed written consent

Exclusion Criteria:

* Diabetes at booking
* Presence of contra-indication to metformin(renal, liver, heart failure)
* moving out of study area for pregnancy management
* Participants who suffer with hyperemesis
* Participants who are 18 years and below
* Participants with significantly raised creatinine
* Participants with high alcohol intake

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2010-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Birth Weight centile (z-score) | At Birth

SECONDARY OUTCOMES:
Maternal Weight gain | Weight at recruitment and at end of pregnancy
Development of Gestational Diabetes | 28 weeks of pregnancy
  A Glucose Tolerance Test would be conducted at 28 wks of pregnancy to diagonose diabetes
Development of hypertension/Preeclampsia | Throughout pregnancy
  Blood Pressure and urinary proteins would be monitored at each visit to diagonose hypertension/Preeclampsia
Caesarian Section | delivery
Postpartum haemorrhage | Delivery
Neonatal Hypoglycemia | within 2 hours after birth and immediate post birth
  Blood glucose is checked within 2 hours after birth and before each feeding until consecutive glucose values of 2.6 mmol per liter (46.8 mg per deciliter) or greater were achieved.
  Neonatal hypoglycemia was defined as 2 capillary plasma glucose levels< 2.6 mmol/l at least 30 minutes apart.
Prematurity | Delivery
  Born < 37 weeks gestation
Hyperbilirubinemia | at birth and after
  Hyperbilirubinemia requiring phototherapy
Polycythaemia | At birth
  Cord blood hematocrit > 0.6
Respiratory Distress | At birth and within 24 hours
  4 or more hours of respiratory suppory or oxygen with associated diagnosis
Macrosomia/Large for Gestational Age | At birth
  Birth weight>90th centile based on appropriate growth standards
Birth Trauma | At birth
  Shoulder dystocia, brachial plexus injury
Apgar score <6 | 5 minutes after birth
Admission to level 2 or greater neonatal unit | at birth and immediately after
  If yes, then length of stay
Stillbirth/Intrauterine deaths | Throughout pregnancy
2nd trimester miscarriages | in 2nd trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mr Hassan Shehata, MD MRCOG, Principal Investigator — Epsom and St Helier University Hospitals NHS Trust; Dr Steve Hyer, MD, FRCP, Study Director — Epsom and St Helier University Hospitals NHS Trust; Prof Kypros Nicolaides, PhD, MRCOG, Principal Investigator — King's College London; Dr Jyoti Balani, MD, Principal Investigator — Epsom and St Helier University Hospitals NHS Trust; Dr Ranjit Akolekar, Principal Investigator — Medway Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - Medway Hospital NHS Trust, Gillingham, Kent
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton, Surrey
  - Kings College, London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balani J, Hyer SL, Rodin DA, Shehata H. Pregnancy outcomes in women with gestational diabetes treated with metformin or insulin: a case-control study. Diabet Med. 2009 Aug;26(8):798-802. doi: 10.1111/j.1464-5491.2009.02780.x. PMID 19709150
- [Background] Glueck CJ, Goldenberg N, Wang P, Loftspring M, Sherman A. Metformin during pregnancy reduces insulin, insulin resistance, insulin secretion, weight, testosterone and development of gestational diabetes: prospective longitudinal assessment of women with polycystic ovary syndrome from preconception throughout pregnancy. Hum Reprod. 2004 Mar;19(3):510-21. doi: 10.1093/humrep/deh109. Epub 2004 Jan 29. PMID 14998944
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Galtier-Dereure F, Boegner C, Bringer J. Obesity and pregnancy: complications and cost. Am J Clin Nutr. 2000 May;71(5 Suppl):1242S-8S. doi: 10.1093/ajcn/71.5.1242s. PMID 10799397
- [Derived] Syngelaki A, Nicolaides KH, Balani J, Hyer S, Akolekar R, Kotecha R, Pastides A, Shehata H. Metformin versus Placebo in Obese Pregnant Women without Diabetes Mellitus. N Engl J Med. 2016 Feb 4;374(5):434-43. doi: 10.1056/NEJMoa1509819. PMID 26840133